CLINICAL TRIAL: NCT05252078
Title: An Open, Single Arm, Multicenter, Exploratory Phase II Clinical Trial of Anlotinib Hydrochloride Capsules Combined With TQB2450 Injection in Esophageal Squamous Cell Carcinoma Patients as Postoperative Adjuvant Therapy
Brief Title: Anlotinib Hydrochloride Capsules Combined With TQB2450 Injection in Esophageal Squamous Cell Carcinoma Patients
Acronym: ALTER-E005
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021ky222
Record Dates: First submitted 2022-01-22; First posted 2022-02-23 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms; Esophageal Diseases; Gastrointestinal Neoplasms; Gastrointestinal Diseases; Digestive System Neoplasms; Digestive System Diseases; Neoplasms by Site; Neoplasms by Histologic Type; Neoplasms, Squamous Cell; Carcinoma, Squamous Cell
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms; Esophageal Diseases; Gastrointestinal Neoplasms; Gastrointestinal Diseases; Digestive System Neoplasms; Digestive System Diseases; Neoplasms by Site; Neoplasms by Histologic Type; Neoplasms, Squamous Cell; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib (Experimental): Patients in the study group will receive the following treatment:
  21 days as a treatment cycle, Anlotinib 12 mg/day, Orally (D1-D14); TQB 2450 1200 mg, iv (D1).
  If anlotinib is not tolerated, the dose can be reduced to 10mg or 8mg, until un-tolerable toxicity again.
  Interventions: Drug: Anlotinib hydrochloride; Drug: TQB2450

INTERVENTIONS:
Drug: Anlotinib hydrochloride — Anlotinib Hydrochloride is a capsule in the form of 8 mg ,10 mg and 12 mg, orally, once daily, 2 weeks on/1 week off.
Drug: TQB2450 — TQB2450 is an injection in the form of 600 mg; 1200 mg, iv, D1.

SUMMARY:
This is an Open, Single Arm, Exploratory and Phase II Clinical Trial of Anlotinib Hydrochloride Capsules Combined With TQB2450 Injection in Esophageal Squamous Cell Carcinoma (ESCC) Patients as Postoperative Adjuvant Therapy. In order to observe and evaluate the efficacy and safety of Anlotinib Hydrochloride Capsules combined with TQB2450 Injection in treatment of patients with ESCC. The primary endpoint is disease free survival (DFS).

DETAILED DESCRIPTION:
This is an Open, Single Arm, Exploratory and Phase II Clinical Trial of Anlotinib Hydrochloride Capsules Combined With TQB2450 Injection in Esophageal Squamous Cell Carcinoma (ESCC) Patients as Postoperative Adjuvant Therapy. In order to observe and evaluate the efficacy and safety of Anlotinib Hydrochloride Capsules combined with TQB2450 Injection in treatment of patients with Esophageal Squamous Cell Carcinoma (ESCC). Primary Efficacy Endpoint: Disease Free Survival (DFS) (According to RECIST Version 1.1), Secondary Efficacy Endpoints:1-year DFS rate, 3-year DFS rate, 1-year Overall Survival (OS) rate, 3-year OS rate, and Safety. Safety and tolerance will be evaluated by incidence, severity and outcomes of AEs and categorized by severity in accordance with the NCI CTC AE Version 5.0.

ELIGIBILITY:
Inclusion Criteria:

* Subjects volunteered to join the study, signed informed consent, good compliance, with follow-up.
* ≥ 18 years old.
* ECOG performance status of 0-1
* Patients with esophageal squamous cell carcinoma pathologically diagnosed as T1-2N1-3M0 or T3-4NanyM0.
* Patients received radical (R0) resection of squamous cell carcinoma with no recurrence in imaging examination within 6-12 weeks after surgery, and need adjuvant therapy assessed by the researchers.
* Laboratory tests must be met:
* Neutrophils count =/> 1.5 x 109/L, platelets count =/> 75 x 109/L, Hb =/> 90 g/L, WBC =/> 3 x 109/L.
* total bilirubin =/< 1.5 x ULN, ALT and AST =/< 2.5 x ULN.
* Creatinine =/< 1.5 x ULN.
* APTT, INR, PT =/< 1.5 x ULN.
* TSH =/< ULN.
* Myocardial enzymes in the normal range.
* LVEF =/> 50%.

Exclusion Criteria:

* Patients received other antitumor adjuvant therapy after surgical resection.
* Concurrent malignancy (except cured basal cell carcinoma of the skin).
* Patients was diagnosed cervical esophageal carcinoma.
* Patients who have received prior targeted therapy (anti-VEGF/VEGFR) or immunity therapy (anti-PD-1/PD-L1/CTLA-4).
* Patients who are allergic to other monoclonal antibodies.
* Patients with a history of immunodeficiency (or active autoimmue disease), or other acquired congenital immunodeficiency diseases.
* Immunosuppressant, systemic, or absorbable local hormone therapy (> 10mg/ day of prednisone or other equivalent hormone) is required for immunosuppression and continued within 2 weeks of initial administration.
* Patients with multiple factors affecting oral administration.
* Uncontrolled pleural effusion, pericardial effusion or ascites that requires repeated drainage.
* With bleeding tendency. Patients with any bleeding or bleeding event CTC AE grade 3 in the 4 weeks prior to initial administration. The presence of digestive diseases or active bleeding of unresected tumors, or other conditions that the investigator determined which could lead to gastrointestinal bleeding or perforation.
* Active or untreated CNS metastases as determined by CT or magnetic resonance imaging (MRI) evaluation during screening and prior radiographic assessments.
* Patients with hypertension who could not be well controlled by antihypertensive drugs (systolic blood pressure > 160 mmHg, diastolic blood pressure > 100 mmHg).
* Patients with myocardial infarction, myocardial ischemia, arrhythmias with poor control (including QTC interval male > 450 ms, female> 470 ms) and cardiac insufficiency of grade II according to NYHA standard.
* Active or uncontrolled severe infection (≥ CTC AE Grade 2 infection).
* HIV test positive.
* Proteinuria =/>2+ and confirmed 24-hour urinary protein quantification > 1.0 g.
* Vaccination with prophylactic or attenuated vaccine within 4 weeks prior to initial administration.
* According to the investigators' judgment, there are factors that endanger patient or prevent patients from completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
DFS | DFS was defined as the time from the day patients received first dose of treatment regimen until the date of first documented recurrence or death from any cause, whichever come first, assessed up to 96 months.
  Disease Free Survival

SECONDARY OUTCOMES:
1-year DFS rate | 1-year DFS rate was disease-free survival rate at the time since patients received first dose of treatment regimen for one year.
  One year Disease Free Survival rate
3-year DFS rate | 3-year DFS rate was disease-free survival rate at the time since patients received first dose of treatment regimen for 3 years.
  Three year Disease Free Survival rate
1-year OS rate | 1-year OS rate was overall survival rate at the time since patients received first dose of treatment regimen for one year.
  One year Overall Survival rate
3-year OS rate | 3-year OS rate was overall survival rate at the time since patients received first dose of treatment regimen for 3 years.
  Three year Overall Survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Changying Guo, PhD, Principal Investigator — Jiangxi Provincial Cancer Hospital
Locations (1):
- Jiangxi Cancer Hospital, Nanchang, Jiangxi, China